CLINICAL TRIAL: NCT02763878
Title: Uncut Roux-en-y Anastomosis Reduce Postoperative Complication and Improve Nutritional Status After Distal Gastrectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CSGC-002
Record Dates: First submitted 2016-02-05; First posted 2016-05-05 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-05

CONDITIONS: Nutrition Disorders; Postoperative Complications
Keywords: Uncut Roux-en-Y; Billroth II anastomosis; Distal gastric cancer; Nutrition status; Postoperative complications
MeSH Terms: conditions — Nutrition Disorders; Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- uncut Roux-en-Y anastomosis (Experimental): After distal gastrectomy, duodenal stump closure, side to side anastomosis was underwent on the remnant stomach and jejunum,which was 25cm from Treitz ligament. Then underwent side to side anastomosis between jejunum about 35cm distance from gastrojejunostomy and jejunum about 5cm from Triez ligament . close the intestinal cavity on the input less than 5cm distance from the loop gastrojejunostomy anastomosis by using uncut Closure devices
  Interventions: Procedure: Uncut Roux-en-Y anastomosis
- Billroth II anastomosis (Sham Comparator): After distal gastrectomy, duodenal stump closure, the investigators first underwent remnant stomach and upper jejunum side anastomosis. Then choose the jejunum about 25cm from Treitz ligament, premenstrual colon using a disposable cutting closure (or tubular stapling) in the rear wall of the stomach and jejunum anastomosis, common opening was closed with the (barbed wire) hand-stitched. After that, steps were same with the group A.
  Interventions: Procedure: Billroth II anastomosis

INTERVENTIONS:
Procedure: Uncut Roux-en-Y anastomosis — Uncut Closure devices would be used to close the intestinal cavity on the input less than 5cm distance from the loop gastrojejunostomy anastomosis.
  Arms: uncut Roux-en-Y anastomosis
Procedure: Billroth II anastomosis — Typical Billroth II anastomosis would be made after the Distal gastrectomy.
  Arms: Billroth II anastomosis

SUMMARY:
The investigators intend to conduct multi-center randomized controlled study to find if Uncut Roux-en-Y anastomosis to the distal gastric cancer patients after radical D2 can reduce the long-term complications, affect the quality of life, and improve the prognosis, comparing to Billroth II anastomosis.

DETAILED DESCRIPTION:
Gastric cancer is still one of the most common malignant tumors, and gastric antrum cancer is still common. Radical surgery is the only way to treat gastric antrum cancer, surgical procedures and reconstruction are closely related with the prognosis and quality of life, the choice is crucial. Gastrojejunostomy after distal gastrectomy may affect the quality of radical surgery, and postoperative diet, nutritional status and quality of life. More and more centers tend to choose Billroth II anastomosis, but patients prone to have a variety of complications, including reflux gastritis and bile reflux, malnutrition, seriously affecting the quality of life and so on. According to preliminary pilot study found that, uncut Roux-en-Y anastomosis way can keep the continuity of nerve-muscle function of the reconstruction of digestive tract, and closes the input in order to reduce the incidence of reflux, for improving the nutritional status and reducing complications and improve quality of life. Therefore, the investigators intend to conduct multi-center randomized controlled study to find if Uncut Roux-en-Y anastomosis to the distal gastric cancer patients after radical D2 can reduce the long-term complications, affect the quality of life, and improve the prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. pathological diagnosed as the gastric carcinoma, the possibility of removal by the surgeon and imaging physician assessment.
2. no previous history of other malignancies combined.
3. patients have signed informed consent;
4. aged 18 to 80 years old, male or female patients;
5. cardiopulmonary, liver and kidney function was normal, ECOG physical status score of 0 to 1 (see Appendix);
6. the clinician determine the patient does not need emergency surgery;

Exclusion Criteria:

1. pregnant or lactating women;
2. the liver, lung, bone, and other distant metastasis;
3. supraclavicular lymph nodes, pelvic or ovarian species, peritoneal dissemination, etc;
4. a large number of ascites, cachexia;
5. suffering from other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, poorly controlled hypertension merger, diabetes patients;
6. or mental illness;
7. 4 weeks prior to enrollment participated or are participating in other clinical trials of patients;
8. had undergone surgery, and its influence has not been eliminated in the patient;
9. of the stomach or esophagus history of malignancy, including stromal tumor, sarcoma, lymphoma, carcinoid;
10. patients with active infection (infection causing fever above 38 ℃);
11. patients with poor compliance or researchers consider poor patient compliance;
12. There are other clinical researchers believe that the laboratory the patient should not participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 832 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related gastrointestinal and gastroesophageal reflux as assessed by The Los Angeles and Savary-Miller systems for grading esophagitis | 0-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Sheng Peng, Ph.D, Principal Investigator — The sixth affliated hospital of Sun Yat-sen University
Locations (1):
- The sixth affliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The investigators would like to share the data to the Participating units.

REFERENCES:
- [Result] Yun SC, Choi HJ, Park JY, Kim YJ. Total laparoscopic uncut Roux-en-Y gastrojejunostomy after distal gastrectomy. Am Surg. 2014 Feb;80(2):E51-3. No abstract available. PMID 24480200
- [Result] Ahn SH, Son SY, Lee CM, Jung DH, Park do J, Kim HH. Intracorporeal uncut Roux-en-Y gastrojejunostomy reconstruction in pure single-incision laparoscopic distal gastrectomy for early gastric cancer: unaided stapling closure. J Am Coll Surg. 2014 Jan;218(1):e17-21. doi: 10.1016/j.jamcollsurg.2013.09.009. Epub 2013 Nov 23. No abstract available. PMID 24280449
- [Result] Mon RA, Cullen JJ. Standard Roux-en-Y gastrojejunostomy vs. "uncut" Roux-en-Y gastrojejunostomy: a matched cohort study. J Gastrointest Surg. 2000 May-Jun;4(3):298-303. doi: 10.1016/s1091-255x(00)80079-7. PMID 10769093
- [Derived] Cai Z, Mu M, Ma Q, Liu C, Jiang Z, Liu B, Ji G, Zhang B. Uncut Roux-en-Y reconstruction after distal gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2024 Feb 29;2(2):CD015014. doi: 10.1002/14651858.CD015014.pub2. PMID 38421211
- [Derived] Chen S, Chen DW, Chen XJ, Lin YJ, Xiang J, Peng JS. Postoperative complications and nutritional status between uncut Roux-en-Y anastomosis and Billroth II anastomosis after D2 distal gastrectomy: a study protocol for a multicenter randomized controlled trial. Trials. 2019 Jul 12;20(1):428. doi: 10.1186/s13063-019-3531-0. PMID 31300019